CLINICAL TRIAL: NCT02652650
Title: A Phase 1, Open-label Study in Healthy Female Subjects to Investigate the Effect of JNJ-63623872 at Steady-state on the Steady-state Pharmacokinetics of Ethinylestradiol and Norethindrone
Brief Title: A Study to Investigate the Effect of JNJ-63623872 at Steady-state on the Steady-state Pharmacokinetics of Ethinylestradiol and Norethindrone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR108093; 63623872FLZ1009 (Other: Janssen Research & Development, LLC); 2015-000639-34 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Healthy; JNJ-63623872; Ethinylestradiol; Norethindrone
MeSH Terms: interventions — Ethinyl Estradiol; Norethindrone; pimodivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ethinylestradiol/Norethindrone (Experimental): During the first oral contraceptive (OC) cycle participants will receive ethinylestradiol/norethindrone 35 microgram (mcg)/1 milligram (mg) alone once daily (qd) for 21 days on Days 1 to 21 (Cycle I: lead-in). During the second OC cycle (from Day 29 to Day 56), participants will receive ethinylestradiol/norethindrone 35 mcg/1 mg alone qd for 21 days on Days 29 to 49 (Cycle II: OC alone, reference). During the third OC cycle (from Day 57 to Day 84), participants will receive ethinylestradiol/norethindrone 35 mcg/1 mg qd for 21 days on Days 57 to 77 and in addition JNJ-63623872, 600 mg twice daily (bid) for 5 days on Days 73 to 77 (Cycle III: OC plus JNJ-63623872, test).
  Interventions: Drug: Ethinylestradiol; Drug: Norethindrone; Drug: JNJ-63623872

INTERVENTIONS:
Drug: Ethinylestradiol — Participants will receive 35 microgram (mcg) alone once daily (qd) for 21 days on Days 1 to 21 (Cycle I: lead-in) during first OC cycle; Days 29 to 49 (Cycle II: OC alone, reference) during the second OC cycle and Days 57 to 77 during third OC cycle.
Drug: Norethindrone — Participants will receive 1 milligram (mg) alone once daily (qd) for 21 days on Days 1 to 21 (Cycle I: lead-in) during first OC cycle; Days 29 to 49 (Cycle II: OC alone, reference) during the second OC cycle and Days 57 to 77 during third OC cycle.
Drug: JNJ-63623872 — Participants will receive 600 mg twice daily (bid) for 5 days on Days 73 to 77 (Cycle III: OC plus JNJ-63623872, test) during third OC cycle under fed conditions.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state concentrations of JNJ-63623872 on the steady-state pharmacokinetics of ethinylestradiol and norethindrone in healthy female participants.

DETAILED DESCRIPTION:
This is a Phase 1 and open-label study. The study consists of Screening Phase (less than or equal to (<=) 28 days before Day 1), Treatment Phase (Day 1 up to Day 78) and Follow up Phase (10 to 14 days after last study drug intake or, if an adverse event occurs, 30 to 35 days after last study drug intake). Treatment phase will consist of three Oral Contraceptive (OC) cycles (each cycle consists of 21 days of ethinylestradiol/norethindrone followed by 7 pill-free days). The duration of the treatment phase, including the OC-free period of Cycles I and II, will be 78 days. Blood samples will be collected for measurement of pharmacokinetic (Pk) parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing and able to adhere to the prohibitions and restrictions specified in the protocol
* Participants must, if heterosexually active with a partner who is not vasectomized (confirmed sterile), be practicing an effective method of contraception before entry and agree to continue to use two effective methods of contraception throughout the study and for at least 30 days after receiving the last intake of oral contraceptive (OC) plus JNJ-63623872 on Day 77
* Participants must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 of Cycle I
* Participants must agree not to donate eggs (ova, oocytes) during the study and for at least 90 days after receiving the last intake of OC plus JNJ-63623872 on Day 77
* Participants must have a Body Mass Index (BMI); between 18.0 and 30.0 kilogram per square meter (kg/m^2) (extremes included)

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* At screening, participants with one or more of the laboratory abnormalities specified in the protocol as defined by the World Health Organization (WHO) Toxicity Grading Scale
* Participant with a past history of heart arrhythmias (extrasystole, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticarial
* Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of JNJ-63623872 | Post-dose on Days 75 and 76 of Cycle III
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing Interval.
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing Interval.
Observed Analyte Concentration at 12 Hours Post Dosing (C12h) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  C12h is the observed analyte concentration at 12 hours post dosing.
Minimum Observed Analyte Concentration (Cmin) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  Cmin is the minimum observed analyte concentration.
Maximum Observed Analyte Concentration (Cmax) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  Cmax is the maximum observed analyte concentration.
Time To Reach The Maximum Observed Analyte Concentration (Tmax) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  Tmax is the actual sampling time to reach the maximum observed analyte concentration.
Area Under the Analyte Concentration versus Time Curve (AUC) From Time of Administration up to 12 Hours Post Dosing (AUC12h) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  AUC12h is the area under the analyte concentration versus time curve (AUC) from time of administration up to 12 hours post dosing.
Average Steady-State Plasma Concentration (Cavg) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  Cavg is the average steady-state plasma concentration.
Percentage Fluctuation (FI) of JNJ-63623872 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle II
  FI is the percentage fluctuation(variation between maximum and minimum concentration at steady-state), calculated as: 100 multiplied ([Cmax - Cmin] / Cavg).
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of Ethinylestradiol | Post-dose on Days 47 and 48 of Cycle II; post-dose on Days 75 and 76 of Cycle III
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing Interval.
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of Norethindrone | Post-dose on Days 47 and 48 of Cycle II; post-dose on Days 75 and 76 of Cycle III
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing Interval.
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing Interval.
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing Interval.
Observed Analyte Concentration at 24 Hours Post Dosing (C24h) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  C24h is the observed analyte concentration at 24 hours post dosing.
Observed Analyte Concentration at 24 Hours Post Dosing (C24h) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  C24h is the observed analyte concentration at 24 hours post dosing.
Minimum Observed Analyte Concentration (Cmin) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Cmin is the minimum observed analyte concentration.
Minimum Observed Analyte Concentration (Cmin) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Cmin is the minimum observed analyte concentration.
Maximum Observed Analyte Concentration (Cmax) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Cmax is the maximum observed analyte concentration.
Maximum Observed Analyte Concentration (Cmax) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Cmax is the maximum observed analyte concentration.
Time To Reach The Maximum Observed Analyte Concentration (Tmax) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Tmax is the actual sampling time to reach the maximum observed analyte concentration.
Time To Reach The Maximum Observed Analyte Concentration (Tmax) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Tmax is the actual sampling time to reach the maximum observed analyte concentration.
Area Under the Analyte Concentration versus Time Curve (auc) From Time of Administration up to 24 Hours Post Dosing (AUC24h) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  AUC24h is the area under the analyte concentration versus time curve (AUC) from time of administration up to 24 hours post dosing.
Area Under the Analyte Concentration versus Time Curve (auc) From Time of Administration up to 24 Hours Post Dosing (AUC24h) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  AUC24h is the area under the analyte concentration versus time curve (AUC) from time of administration up to 24 hours post dosing.
Average Steady-State Plasma Concentration (Cavg) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Cavg average steady-state plasma concentration.
Average Steady-State Plasma Concentration (Cavg) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Cavg average steady-state plasma concentration.
Percentage Fluctuation (FI) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  FI is the percentage fluctuation(variation between maximum and minimum concentration at steady-state), calculated as: 100 multiplied ([Cmax - Cmin] / Cavg).
Percentage Fluctuation (FI) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  FI is the percentage fluctuation(variation between maximum and minimum concentration at steady-state), calculated as: 100 multiplied ([Cmax - Cmin] / Cavg).
Ratio of Individual Cmax Values Between Test and Reference Treatment (Ratio Cmax, test/ref) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Ratio Cmax, test/ref is the ratio of individual Cmax values between test and reference treatment of ethinylestradiol.
Ratio of Individual Cmax Values Between Test and Reference Treatment (Ratio Cmax, test/ref) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Ratio Cmax, test/ref is the ratio of individual Cmax values between test and reference treatment of Norethindrone.
Ratio of Individual AUC24h Values Between Test and Reference Treatment (Ratio AUC24h, test/ref) of Ethinylestradiol | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Ratio AUC24h, test/ref is the ratio of individual AUC24h values between test and reference treatment of Ethinylestradiol.
Ratio of Individual AUC24h Values Between Test and Reference Treatment (Ratio AUC24h, test/ref) of Norethindrone | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 49 of Cycle II; Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 9 and 12 hours post-dose on Day 77 of Cycle III
  Ratio AUC24h, test/ref is the ratio of individual AUC24h values between test and reference treatment of Norethindrone.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium